CLINICAL TRIAL: NCT05315947
Title: A Single-Dose, Open-Label, Randomized, 2-Way Cross-Over Study to Assess the Bioequivalence Between Brivaracetam Tablet and Dry Syrup in Healthy Male Japanese Study Participants
Brief Title: A Study to Assess the Bioequivalence Between Brivaracetam Tablet and Dry Syrup in Healthy Male Japanese Study Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EP0110
Record Dates: First submitted 2022-03-14; First posted 2022-04-07 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: Healthy Study Participants
Keywords: brivaracetam; Healthy Study Participants; Phase 1; BRV
MeSH Terms: interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A-B (Experimental): Study participants randomized to this arm will receive a single dose of brivaracetam tablet (Treatment A) as reference and single dose of brivaracetam dry syrup (Treatment B) as test in the treatment sequence A-B at pre-specified timepoints.
  Interventions: Drug: brivaracetam
- Treatment B-A (Experimental): Study participants randomized to this arm will receive a single dose of brivaracetam tablet (Treatment A) as reference and single dose of brivaracetam dry syrup (Treatment B) as test in the treatment sequence B-A at pre-specified timepoints.
  Interventions: Drug: brivaracetam

INTERVENTIONS:
Drug: brivaracetam — Study participants will receive a single-dose of brivaractam tablet (reference - Treatment A) administered orally.
  Other Names: BRV; Briviact
Drug: brivaracetam — Study participants will receive a single-dose of brivaractam dry syrup (test - Treatment B) administered orally.
  Other Names: BRV; Briviact

SUMMARY:
The purpose of the study is to demonstrate the bioequivalence between the BRV tablet and BRV as dry syrup after a single oral dose in healthy Japanese male study participants.

ELIGIBILITY:
Inclusion criteria:

* Study participant must be between 20 to 50 years of age (inclusive) at the time of signing the Informed Consent Form (ICF)
* Study participant is overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Study participant is of Japanese descent as evidenced by appearance and verbal confirmation of familial heritage (a study participant has all 4 Japanese grandparents born in Japan)

Exclusion criteria:

* Study participant has used other drugs, including over-the-counter medications, herbal/traditional medicines, or dietary supplements (excluding medicines for external use),with the exception of paracetamol, within 14 days before first administration of IMP or has received a coronavirus disease 2019 (COVID-19) vaccine within 7 days of initiating IMP
* Study participant has used hepatic enzyme-inducing drugs (eg, glucocorticoids, phenobarbital, isoniazid, phenytoin, rifampicin) within 2 months before the first administration of Investigational Medicinal Product (IMP)
* Study participant has a positive result for hepatitis B surface antigen, hepatitis C virus antibody test, human immunodeficiency virus antibody test, or syphilis at Screening Visit
* Study participant has donated blood or plasma or has experienced blood loss ≥400 mL within 90 days, ≥200 mL within 30 days, or has donated any blood or plasma within 14 days before first administration of IMP
* Study participant is a current smoker or has used nicotine-containing products (eg, tobacco, patches, gum) within 30 days before the first administration of IMP
* Consumption of more than 600 mg of caffeine/day (1 cup of coffee contains approximately 100mg of caffeine, 1 cup of tea approximately 30 mg, and 1 glass of cola approximately 20 mg)

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- EP0110 1, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

REFERENCES:
- See also: Product Information — https://www.briviact.com/briviact-PI.pdf?v=1479491757
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in April 2022 and concluded in May 2022.
Pre-assignment Details: The Participant Flow refers to the Randomized Set.
Groups:
- Treatment A-B (Sequence: BRV Tablet - BRV Dry Syrup): Participants randomized to this arm first received a single dose of brivaracetam (BRV) 50 milligrams (mg) tablet (reference), administered orally, in the morning under fasting conditions on Day 1 of Dosing Period 1. After a washout period of 7 to 10 days, participants received a single dose of BRV 50 mg as dry syrup (test), administered orally, in the morning under fasting conditions on Day 1 of Dosing Period 2. Both dosing periods were of 4 days, each with a single administration on Day 1 of each Dosing Period.
- Treatment B-A (Sequence: BRV Dry Syrup - BRV Tablet): Participants randomized to this arm first received a single dose of BRV 50 mg as dry syrup (test), administered orally, in the morning under fasting conditions on Day 1 of Dosing Period 1. After a washout period of 7 to 10 days, participants received a single dose of BRV 50 mg tablet (reference), administered orally, in the morning under fasting conditions on Day 1 of Dosing Period 2. Both dosing periods were of 4 days, each with a single administration on Day 1 of each Dosing Period.
Period: Overall Study
Arm/Group | Treatment A-B (Sequence: BRV Tablet - BRV Dry Syrup) | Treatment B-A (Sequence: BRV Dry Syrup - BRV Tablet)
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS) which consisted of all randomized study participants who received at least 1 dose of the investigational medicinal product (IMP).
Groups:
- BRV (All Participants): All participants received a single dose of either BRV 50 mg tablet or BRV 50 mg as dry syrup, orally, in the morning under fasting conditions on Day 1 of Dosing Period 1. After a washout period of 7 to 10 days, all participants received a single dose of either BRV 50 mg tablet or BRV 50 mg as dry syrup, orally, in the morning under fasting conditions on Day 1 of Dosing Period 2. Each dosing period is of 4 days, with a single administration on Day 1 of Dosing Period.
Arm/Group | BRV (All Participants)
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) for a Single Dose of Brivaracetam
Description: Cmax is the maximum plasma concentration of brivaracetam.
Time Frame: Blood samples for this analysis were collected on Predose (Day 1), 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose
Population: Pharmacokinetic Per Protocol Set (PK-PPS) included all randomized study participants who were included in the SS, had no important protocol deviations (IPDs) that were considered to impact the data validity for analysis of the primary study objective, and had a sufficient number of bioanalytical assessments to calculate reliable estimates for the primary pharmacokinetic parameters for both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Groups:
- BRV Tablet: Participants who received a single administration of BRV 50 mg tablet, under fasting conditions on either Day 1 of Dosing Period 1 or Day 1 of Dosing Period 2 of the study.
- BRV Dry Syrup: Participants who received a single administration of BRV 50 mg as dry syrup, under fasting conditions on either Day 1 of Dosing Period 1 or Day 1 of Dosing Period 2 of the study.
Arm/Group | BRV Tablet | BRV Dry Syrup
Number analyzed (Participants) | 24 | 24
micrograms per milliliter (μg/mL) | 2.286 (24.5) | 1.989 (22.4)
Statistical Analysis 1: Comparison: BRV Tablet vs BRV Dry Syrup; Test type: Equivalence — Bioequivalence between the BRV tablet (reference) and BRV dry syrup (test) formulations were concluded if the 90% CI limits for Cmax was within the 0.80 to 1.25 range; Ratio of Dry Syrup/ Tablet = 0.8700, 90% CI 2-sided [0.7814 to 0.9686]

2. Primary Outcome: Area Under the Curve From 0 to the Time of the Last Quantifiable Concentration (AUC(0-t)) for a Single Dose of Brivaracetam
Description: AUC(0-t) is the area under the curve from time 0 to the time of the last quantifiable concentration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*μg/mL
Arm/Group | BRV Tablet | BRV Dry Syrup
Number analyzed (Participants) | 24 | 24
hours*μg/mL | 17.98 (17.0) | 17.78 (16.2)
Statistical Analysis 1: Comparison: BRV Tablet vs BRV Dry Syrup; Test type: Equivalence — Bioequivalence between the BRV tablet (reference) and BRV dry syrup (test) formulations were concluded if the 90% CI limits for AUC(0-t) was within the 0.80 to 1.25 range; Ratio of Dry Syrup/ Tablet = 0.9890, 90% CI 2-sided [0.9756 to 1.003]

3. Secondary Outcome: Percentage of Participants With at Least One Treatment-emergent Adverse Event (TEAE)
Description: An AE was defined as any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of IMP, whether or not considered related to the IMP. A TEAE was defined as any AE with a start date/time on or after the first dose of IMP or any unresolved event already present before administration of IMP that worsens in intensity following exposure to IMP.
Time Frame: From Baseline to end of Safety Follow-Up, up to 20 days
Population: Safety Set (SS) included all randomized study participants who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | BRV Tablet | BRV Dry Syrup
Number analyzed (Participants) | 24 | 24
percentage of participants | 37.5 | 37.5

4. Secondary Outcome: Percentage of Participants With at Least One Treatment-emergent Serious Adverse Event (SAE)
Description: A TEAE was any AE with a start date/time on or after the first dose of IMP or any unresolved event already present before administration of IMP that worsens in intensity following exposure to IMP. A serious adverse event (SAE) was defined as any untoward medical occurrence that at any dose: Results in death, Is life-threatening, Requires in patient hospitalization or prolongation of existing hospitalization,Is a congenital anomaly or birth defect, Is an infection that requires treatment parenteral antibiotics, Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Baseline to end of Safety Follow-Up, up to 20 days
Population: Safety Set (SS) included all randomized study participants who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | BRV Tablet | BRV Dry Syrup
Number analyzed (Participants) | 24 | 24
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline to end of Safety Follow-Up, up to 20 days
Description: A TEAE was defined as any AE with a start date/time on or after the first dose of IMP or any unresolved event already present before administration of IMP that worsens in intensity following exposure to IMP. Safety Set (SS) included all randomized study participants who received at least 1 dose of the IMP.
Arm/Group | BRV Tablet | BRV Dry Syrup
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 9/24 | 8/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BRV Tablet (N=24) | BRV Dry Syrup (N=24)
Somnolence (Nervous system disorders) | 7 (7) | 6 (6)
Dizziness (Nervous system disorders) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT05315947/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT05315947/SAP_001.pdf